CLINICAL TRIAL: NCT03589924
Title: A Randomized Multicenter, Open, Prospective, Controlled Study-comparison of the Safety of Immediate One-stage Implant Based Breast Reconstruction(IBBR) Versus Two-stage Expander-Implant IBBR Augmented With TiLoop® Bra.
Brief Title: Study to Compare the Safety of Immediate One-stage IBBR With Expander-Implant Two-stage IBBR Augmented With TiLoop® Bra(COSTA)
Acronym: IBBR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiong Wu (Other)
Collaborators: First Hospital of China Medical University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor-Investigator, Jiong Wu, professor, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBCSG-040
Record Dates: First submitted 2018-06-16; First posted 2018-07-18 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
Keywords: Immediate implant reconstruction; TiLoop® Bra
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients will undergo Skin Sparing Mastectomy(SSM)/Nipple Sparing Mastectomy(NSM) with one-stage or two stage IBBR with TiLoop® Bra.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One step method (Experimental): Immediate implant reconstruction following mastectomy using TiLoop®Bra (one step method) n=225
  Interventions: Procedure: Immediate IBBR+TiLoop®Bra
- Two step method (Active Comparator): Immediate-delayed implant reconstruction following mastectomy using TiLoop®Bra (two step method) n=225
  Interventions: Procedure: Immediate-delayed IBBR+TiLoop®Bra

INTERVENTIONS:
Procedure: Immediate IBBR+TiLoop®Bra — Patients will receive immediate implant reconstruction following mastectomy using TiLoop®Bra
  Arms: One step method
Procedure: Immediate-delayed IBBR+TiLoop®Bra — Patients will receive immediate-delayed implant reconstruction following mastectomy using TiLoop®Bra
  Arms: Two step method

SUMMARY:
This study is the first prospective randomized study assessing the safety and patient-reported outcomes of immediate one-stage IBBR compared with those of two-stage IBBR with TiLoop® Bra.

DETAILED DESCRIPTION:
Studies comparing two-stage implant-based breast reconstruction with immediate one-stage implant-based breast reconstruction have inconsistent results and investigators find that there is a lack of high quality evidence focusing on comparing one-stage and two-stage implant-based breast reconstruction with TiLoop®Bra.

This study is the first prospective randomized study assessing the safety and patient-reported outcomes of immediate one-stage IBBR compared with those of two-stage IBBR with TiLoop® Bra in breast cancer patients.

The hypothesis is that one step method is not inferior to two step method in implant based breast reconstruction following skin-sparing and/or Nipple-sparing mastectomy using TiLoop® Bra.

The current study is a randomized multicenter, open labeled, prospective, controlled study.

Participants were enrolled at six hospitals in different places of China. All participants will undergo Skin Sparing Mastectomy(SSM)/Nipple Sparing Mastectomy(NSM) with one-stage or two stage IBBR with TiLoop® Bra.

Based on earlier experience, investigators calculated that the surgical complication rate was approximately 30 percent in the one-stage group and 25 percent in the two-stage group. Consider a dropout rate of 5%, a total of 450 patients, with 225 in each group, are needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological proven invasive breast cancer or ductal carcinoma in situ;
* Clinical T1-T2 disease with no distant metastasis;
* Patient with clinical N0 status;
* Intent to receive NSM or SSM and implant based breast reconstruction;
* Signed consent to participate.

Exclusion Criteria:

* Patient with severe breast ptosis;
* Patient received ipsilateral breast reduction or enlargement;
* Locally advanced stage patients who received neoadjuvant chemotherapy or hormone therapy;
* Patients enrolled in other clinical trial which may as influence the outcome;
* Patients received neo-adjuvant therapy and will receive radiotherapy.
* History of breast cancer (ipsilateral, i.e. recurrence, or contralateral breast);
* Patients of pregnancy or lactation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of perioperative complications | Start of randomization until 3 months after surgery
  The rate of perioperative complication between the two groups

SECONDARY OUTCOMES:
Quality of life:EORTC QLQ C30 /+ BR23 questionnaire | 18 months after surgery
  EORTC QLQ C30 /+ BR23(EORTC breast cancer-specific quality of life) questionnaire to evaluate quality of life.
  Participants report the extent to which they have experienced those symptoms or problems during the past week. Each of the symptoms or problems is indicated with four extents, including "not at all" for 1 score,"a little" for 2 score, "quit a bit" for 3 score and "very much" for 4 score. A higher score indicated a worse quality of life.
Patient satisfaction:Breast-Q questionnaire | 18 months after surgery
  Breast-Q questionnaire to evaluate patients' satisfaction Using the reconstruction module of BREAST-Q to evaluate patient-reported outcome (PRO) of the surgery.For each subtheme, one or more BREAST-Q scales were developed to examine specific aspects of patient satisfaction.
  Patient responses to each scale's items are transformed through the Q-Score scoring software to provide a total scale score that ranges from 0 to 100. For all BREAST-Q scales, a higher score means greater satisfaction.
Aesthetic score of reconstructed breast | 18 months after surgery
  Harris evaluation system to evaluate patients' breast aesthetic after surgery. Harris evaluation system is a 4-staged subjective evaluation method scored as "excellent," "good," "fair," "poor" .
Additional surgery | 18 months after surgery
  The type of additional surgery following breast reconstruction
Angiopathology-related assessment of Tiloop bra | 18 months after surgery
  The angiopathology-related assessment in immediate-delayed reconstruction group

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Wu, M.D., Principal Investigator — Fudan University
Locations (11):
- China (11):
  - Sun Yat-sen Memorial Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Guangdong Women and Children Hospital, Guangzhou, Guangdong
  - Hebei Cancer Hospital, Shijiazhuang, Hebei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The first hospital of China medical university, Shengyang, Liaoning
  - Liaoning Cancer Hospital & Insitute, Shenyang, Liaoning
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Cancer Hospital/ Institute, Fudan University, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chi W, Zhang Q, Li L, Chen M, Xiu B, Yang B, Wu J. Immediate Breast Reconstruction After Neoadjuvant Chemotherapy: Factors Associated With Surgical Selection and Complications. Ann Plast Surg. 2023 Jul 1;91(1):48-54. doi: 10.1097/SAP.0000000000003574. Epub 2023 May 19. PMID 37216212